CLINICAL TRIAL: NCT04954326
Title: A Multicentre, Phase II Randomized Study, Open-label, With 2-arm Parallel Group, Comparing the Pharmacokinetics of the Liquid and the Lyophilized Formulations of Pegaspargase (S95014) in Treatment of Paediatric Patients With Newly-Diagnosed Acute Lymphoblastic Leukemia (ALL)
Brief Title: A Study Comparing the Blood Levels of Both Pegaspargase (S95014) Formulations (Liquid vs Lyophilized) in the Treatment of Paediatric Patients With Acute Lymphoblastic Leukemia (ALL)
Acronym: ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry); Les Laboratoires Servier (L.L.S), Russia (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL2-95014-002; 2020-004894-29 (EudraCT Number)
Record Dates: First submitted 2021-06-18; First posted 2021-07-08 (Actual); Results first posted 2023-07-05 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Oncology / Haematology; Phase II; Acute Lymphoblastic Leukemia; Parallel group; Pegaspargase; Pharmacokinetics comparability; Lyophilized pegaspargase; Liquid pegaspargase; Pegaspargase formulation; Randomized, open-label
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S95014 lyophilizate (Experimental): Lyophilized S95014 reconstituted will provide 5 mL of extractable volume with the concentration of 750 U/mL. The vial of lyophilized powder (3.750 U/vial) is reconstituted with 5.2 mL of Sterile Water for Injection to obtain a 750 U/mL solution for single use.
  Interventions: Drug: Lyophilized S95014
- S95014 liquid (Active Comparator): Liquid S95014 is provided as 3.750 U per 5 mL solution in a single use vial to obtain a 750 U/mL solution for single use.
  Interventions: Drug: Liquid S95014

INTERVENTIONS:
Drug: Lyophilized S95014 — Lyophilized S95014 will be intravenously administered over 1 hour at the dose of 2500 U/m2 at Day 3 of the induction phase.
  Patients will receive other backbone chemotherapy agents as per ALL-MB 2015 protocol.
  Arms: S95014 lyophilizate
Drug: Liquid S95014 — Liquid S95014 will be intravenously administered over 1 hour at the dose of 2500 U/m2 at Day 3 of the induction phase.
  Patients will receive other backbone chemotherapy agents as per ALL-MB 2015 protocol.
  Arms: S95014 liquid

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (PK) of both lyophilized and liquid S95014 formulations during the induction phase after a single IV dose in newly diagnosed paediatric patients with ALL

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 to < 18 years
* Patients with cytologically confirmed and documented newly diagnosed ALL according to National Comprehensive Cancer Network guidelines 2020 (see Appendix 2), excluding B-cell Burkitt ALL
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2 (see Appendix 3)
* Highly effective contraception method
* Signed informed consent and assent, when appropriate

Non-inclusion Criteria:

* Unlikely to cooperate in the study
* Pregnant and lactating women
* Participation in another interventional study at the same time; participation in non-interventional registries or epidemiological studies is allowed
* Participant already enrolled in the study (informed consent signed)
* Women of childbearing potential tested positive in a serum pregnancy test within 7 days prior to the treatment period
* Inadequate hepatic function (bilirubin > 1.5 times upper limit of normal (ULN), transaminases > 5x ULN)
* Inadequate renal function defined as serum creatinine > 1.5 x ULN
* Prior treatment with chemotherapy or radiotherapy (except steroids and intrathecal therapy)
* Prior surgery or bone marrow transplant related to the studied disease
* Down Syndrome
* Psychiatric illness/social situation that would limit compliance with study requirements
* Known history of pancreatitis
* Known history of significant liver disease
* Known carriers of HIV antibodies
* Significant laboratory abnormality likely to jeopardize the patients' safety or to interfere with the conduct of the study, in the investigator's opinion
* Pre-existing known coagulopathy (e.g. haemophilia and known protein S deficiency)
* History of previous or concurrent malignancy
* History of sensitivity to polyethylene glycol (PEG) or PEG-based drugs
* Severe or uncontrolled active acute or chronic infection
* Uncontrolled intercurrent illness including life-threatening acute tumor lysis syndrome (e.g. with renal failure), symptomatic congestive heart failure, cardiac arrhythmia

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Isaakovich Karachunskiy, PhD, Principal Investigator — Director of Institute of Oncology, Radiology and Nuclear Medicine. Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology.
Locations (6):
- Russia (6):
  - Regional Children Clinical Hospital, Chelyabinsk
  - Children Regional Clinical Hospital, Krasnodar
  - Russian Children Clinical Hospital, Moscow
  - Regional Children Hospital, Nizhny Novgorod
  - V.A. Almazov National Medical Research Center, Saint Petersburg
  - Regional Children Clinical Hospital, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com
- Available data/document: Study Protocol — https://clinicaltrials.servier.com
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a sceening period (from Day-14 to Day-1) to check the eligibility of the patient in the study
Groups:
- S95014 Lyophilizate: Lyophilized S95014 reconstituted will provide 5 mL of extractable volume with the concentration of 750 U/mL. The vial of lyophilized powder (3.750 U/vial) is reconstituted with 5.2 mL of Sterile Water for Injection to obtain a 750 U/mL solution for single use.
  Lyophilized S95014: Lyophilized S95014 will be intravenously administered over 1 hour at the dose of 2500 U/m2 at Day 3 of the induction phase.
  Patients will receive other backbone chemotherapy agents as per ALL-MB 2015 protocol.
- S95014 Liquid: Liquid S95014 is provided as 3.750 U per 5 mL solution in a single use vial to obtain a 750 U/mL solution for single use.
  Liquid S95014: Liquid S95014 will be intravenously administered over 1 hour at the dose of 2500 U/m2 at Day 3 of the induction phase.
  Patients will receive other backbone chemotherapy agents as per ALL-MB 2015 protocol.
Period: Overall Study
Arm/Group | S95014 Lyophilizate | S95014 Liquid
Started | 44 | 45
Completed | 44 (One patient randomized into the lyophilizate group received the liquid formulation in error and was classified according to the treatment actually received. They are counted here as the lyophilizate group, as that is what they were initially randomized into. However for the baseline and statistical measures, they are counted in the liquid group, as that is the drug that they received.) | 41 (The reasons for withdrawals were : two deaths, one protocol violation (patient wrongly included with B-cell Burkit ALL and withdrawn before receiving any IMP), and one physician's decision (patient with allergic reaction after starting the infusion with the IMP).)
Not Completed | 0 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient in the S95014 liquid (LIQ) group was prematurely withdrawn from the study on the day of randomization due to a major deviation/protocol violation (patient with B-cell Burkitt Acute Lymphoblastic Leukemia) and did not receive the study treatment. Another patient who was randomized in the lyophilizate (LYO) group but received the LIQ formulation in error, was analyzed according to the treatment actually received, LIQ, and counted here under LIQ.
Groups:
- Total: Total of all reporting groups
Arm/Group | S95014 Lyophilizate | S95014 Liquid | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43 | 45 | 88
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (4.28) | 5.4 (3.52) | 6.1 (3.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 25 | 42
  Male | 26 | 20 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 44 | 84
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Russia | 43 | 45 | 88

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Measurement
Description: Area Under the Plasma Asparaginase activity - Time curve from Time zero to infinity (AUCinf)
Time Frame: Predose up to 600 hours
Population: The Pharmacokinetic (PK) Analysis Set included the patients who have received at least one dose of IMP and are evaluable for PK analysis : the patients who had enough samples collected to provide interpretable PK results with no deviations that might have affected the PK interpretation (e.g. infusion interrupted for any reason, deviation in the theoretical administered dose > 10%, at least one missing PK sample during the 48 first hours, ≥ 2 missing PK samples after the 48-hour time point).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mU*day/mL
Arm/Group | S95014 Lyophilizate | S95014 Liquid
Number analyzed (Participants) | 41 | 39
mU*day/mL | 362028.656 (33.55) | 352248.907 (31.08)
Statistical Analysis 1: Comparison: S95014 Lyophilizate vs S95014 Liquid; AUCinf was natural log-transformed and analyzed using an analysis of variance (ANOVA) with fixed effect for formulation. The two one-sided tests procedures were performed on the geometric mean ratio (GMR) between test (S95014 lyophilizate) and reference (S95014 liquid formulation) treatments. The 90% confidence interval for the ratio was obtained within the framework of the ANOVA; Test type: Equivalence — The 90% Confidence Interval of the geometric mean ratios of the Lyophilisate compared to the Liquid formulations for AUCinf should be completely contained within the predefined [80.00%-125.00%] equivalence interval; p = 0.05, ANOVA; Geometric Mean Ratio (%) = 102.8, 90% CI 2-sided [91.4 to 115.6]

2. Primary Outcome: Pharmacokinetics Measurement
Description: Maximum observed plasma asparaginase activity (Cmax)
Time Frame: Predose up to 600 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mU/mL
Arm/Group | S95014 Lyophilizate | S95014 Liquid
Number analyzed (Participants) | 41 | 40
mU/mL | 1563.115 (23.11) | 1672.136 (41.91)
Statistical Analysis 1: Comparison: S95014 Lyophilizate vs S95014 Liquid; Cmax was natural log-transformed and analyzed using an analysis of variance (ANOVA) with fixed effect for formulation. The two one-sided tests procedures were performed on the geometric mean ratio (GMR) between test (S95014 lyophilizate) and reference (S95014 liquid formulation) treatments. The 90% confidence interval for the ratio was obtained within the framework of the ANOVA; Test type: Equivalence — The 90% Confidence Interval of the geometric mean ratios of the Lyophilisate compared to the Liquid formulations for Cmax should be completely contained within the predefined [80.00%-125.00%] equivalence interval; p = 0.05, ANOVA; Geometric Mean Ratio (%) = 93.5, 90% CI 2-sided [82.9 to 105.5]

3. Secondary Outcome: Pharmacokinetics Measurements
Description: Observed Plasma Asparaginase Activity 14 days post-dose (Cday 14) of S95014
Time Frame: 14 days post-dose
Population: The PKAS included the patients who have received at least one dose of IMP and are evaluable for PK analysis : the patients who had enough samples collected to provide interpretable PK results with no deviations that might have affected the PK interpretation .
  Cday-14 could not be calculated in one patient (in S95014 liquid group) who had only 3 positive values exceeding the Lower Limit of Quantification
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mU/mL
Arm/Group | S95014 Lyophilizate | S95014 Liquid
Number analyzed (Participants) | 41 | 39
mU/mL | 496.599 (37.96) | 408.655 (80.35)
Statistical Analysis 1: Comparison: S95014 Lyophilizate vs S95014 Liquid; Cday14 was natural log-transformed and analyzed using an analysis of variance (ANOVA) with fixed effect for formulation. The two one-sided tests procedures were performed on the geometric mean ratio (GMR) between test (S95014 lyophilizate) and reference (S95014 liquid formulation) treatments. The 90% confidence interval for the ratio was obtained within the framework of the ANOVA; Test type: Equivalence — The 90% Confidence Interval of the geometric mean ratios of the Lyophilisate compared to the Liquid formulations for Cday14 should be completely contained within the predefined [80.00%-125.00%] equivalence interval; p = 0.05, ANOVA; Geometric Mean Ratio (%) = 121.5, 90% CI 2-sided [98.7 to 149.6]

4. Secondary Outcome: Activity Measurement
Description: Plasma Asparaginase Activity (PAA) of ≥ 0.1 U/mL after the administration of either liquid or lyophilized S95014.
Time Frame: Day 7, 14, 18 and 25 post-dose of either liquid or lyophilized S95014
Population: The analysis on the Plasma Asparaginase Actvity was performed on the Safety Set analysis, defined as the set of all patients who had received at least one dose of S95014 in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | S95014 Lyophilizate | S95014 Liquid
Number analyzed (Participants) | 43 | 45
Participants
  Number of patients who achieved Day 10 Plasma Asparaginase Activity (PAA) ≥ 0.1 U/mL: number analyzed (Participants) | 43 | 44
  Number of patients who achieved Day 10 Plasma Asparaginase Activity (PAA) ≥ 0.1 U/mL | 43 | 43
  Number of patients who achieved Day 17 Plasma Asparaginase Activity (PAA) ≥ 0.1 U/mL: number analyzed (Participants) | 43 | 43
  Number of patients who achieved Day 17 Plasma Asparaginase Activity (PAA) ≥ 0.1 U/mL | 43 | 41
  Number of patients who achieved Day 21 Plasma Asparaginase Activity (PAA) ≥ 0.1 U/mL: number analyzed (Participants) | 42 | 43
  Number of patients who achieved Day 21 Plasma Asparaginase Activity (PAA) ≥ 0.1 U/mL | 41 | 39
  Number of patients who achieved Day 28 Plasma Asparaginase Activity (PAA) ≥ 0.1 U/mL: number analyzed (Participants) | 42 | 43
  Number of patients who achieved Day 28 Plasma Asparaginase Activity (PAA) ≥ 0.1 U/mL | 18 | 6

5. Secondary Outcome: Immunogenicity Measurements
Description: Anti-drug antibodies (ADA) formation against S95014 and anti-PEG with the lyophilized or liquid formulations (positive patients).
Time Frame: Pre-dose, post-dose (sum of 14 and 25 days post-dose)
Population: The immunogenicity analyses were carried out in the Immunogenicity Analysis Set (IAS) which includes all patients who had received at least one dose of IMP and had at least one post-dose sample evaluable for immunogenicity testing.
Measure: Count of Participants; unit: Participants
Arm/Group | S95014 Lyophilizate | S95014 Liquid
Number analyzed (Participants) | 43 | 43
Participants
  Pre-dose: Anti-S95014 Negative/ Anti-PEG Not applicable | 38 | 38
  Pre-dose: Anti-S95014 Positive / Anti-PEG Positive | 2 | 4
  Pre-dose: Anti-S95014 Positive / Anti-PEG Negative | 3 | 1
  Post-dose (sum of 14 and 25 days post-dose): Anti-S95014 Negative/ Anti-PEG Not applicable | 38 | 39
  Post-dose (sum of 14 and 25 days post-dose): Anti-S95014 Positive / Anti-PEG Positive | 2 | 3
  Post-dose (sum of 14 and 25 days post-dose): Anti-S95014 Positive / Anti-PEG Negative | 3 | 1

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected was1,5 month.
Arm/Group | S95014 Lyophilizate | S95014 Liquid
All-Cause Mortality (participants affected / at risk) | 1/43 | 2/45
Serious Adverse Events (participants affected / at risk) | 19/43 | 18/45
Other Adverse Events (participants affected / at risk) | 43/43 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S95014 Lyophilizate (N=43) | S95014 Liquid (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Hypofibrinogenemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 4 (4)
White blood cell count decreased (Investigations) | 4 (4) | 2 (2)
Antithrombin III decreased (Investigations) | 2 (2) | 1 (1)
Blood fibrinogen decreased (Investigations) | 2 (2) | 1 (1)
ALT increased (Investigations) | 1 (1) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Protein S decreased (Investigations) | 1 (1) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Edematous pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis hemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Candida pneumonia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 2 (2)
Catheter site thrombosis (General disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Tonic convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pelvic Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S95014 Lyophilizate (N=43) | S95014 Liquid (N=45)
Blood fibrinogen decreased (Investigations) | 35 (35) | 38 (40)
Antithrombin III decreased (Investigations) | 32 (33) | 32 (32)
Lymphocyte count decreased (Investigations) | 32 (34) | 27 (33)
White blood cell count decreased (Investigations) | 19 (19) | 15 (15)
Leukopenia (Blood and lymphatic system disorders) | 16 (16) | 12 (12)
Alanine aminotransferase increased (Investigations) | 9 (10) | 17 (18)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 16 (17)
Blood bilirubin increased (Investigations) | 13 (14) | 12 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9) | 13 (13)
Protein S decreased (Investigations) | 10 (10) | 9 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (10) | 8 (9)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 10 (10)
Toxic neuropathy (Nervous system disorders) | 11 (11) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 8 (10)
Ammonia increased (Investigations) | 5 (5) | 6 (6)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 7 (7)
Neutropenic colitis (Gastrointestinal disorders) | 6 (6) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 5 (5)
Hypofibrinogenemia (Blood and lymphatic system disorders) | 5 (6) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6)
Platelet count decreased (Investigations) | 4 (4) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 5 (5) | 1 (1)
Blood albumin decreased (Investigations) | 2 (2) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (4)
Hyperbilirubinemia (Hepatobiliary disorders) | 4 (7) | 1 (1)
International normalized ratio increased (Investigations) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Blood urea increased (Investigations) | 3 (4) | 1 (1)
Hemoglobin decreased (Investigations) | 1 (1) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT04954326/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT04954326/SAP_001.pdf